CLINICAL TRIAL: NCT01734603
Title: Randomized, Monocentric and Multidisciplinary Study of the Effects of an Intensive Rehabilitation by Interval Training With Active Recovery in Peripheral Arterial Disease With Claudication
Brief Title: Intensive Rehabilitation in Peripheral Arterial Disease With Claudication: Effects of a Treadmill Training With Active Recovery
Acronym: ARTEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 12
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: Assessment; Rehabilitation; Walking Constant Test; Walking Graded test; Six minute Walking test; Walking Distance
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional rehabilitation program (Active Comparator): conventional rehabilitation program 20 patients are expected in this arm. Patients perform walking treadmill exercises with complete rest.
  Interventions: Procedure: conventional rehabilitation program
- experimental rehabilitation program (Experimental): experimental rehabilitation program 20 patients are expected in this arm. Patients perform walking treadmill exercises with active recovery (no stop walking).
  Interventions: Procedure: experimental rehabilitation program

INTERVENTIONS:
Procedure: experimental rehabilitation program — Duration training = 40 min : 5 cycles of 6 min each Week 1 speed of the walking exercise fixed at 70% of the max walking test's speed done on the initial walking test speed of the walking recovery fixed at 40% Walking slope : 0% Increase of the speed = 0.1 km/h after each training without pain.
  * Week 2 Walking speed = average of the walking speeds done on week 1 Walking slope = 1% Recovery slope = 0% Increase of the slope = 0.5% after each training without pain.
  * Week 3 Walking speed = 70% of the maximal walking test's speed Recovery speed = 40 % of the maximal walking test's speed Slope = average of the slopes done on week 2 Increase of the speed = 0.1 km/h .
  * Week 4 Speeds = average of the walking speeds done on week 3 Walking slope = 1% Recovery slope = 0% Increase of the slope is 0.5% .
  Arms: experimental rehabilitation program
Procedure: conventional rehabilitation program — Duration of the training 40 minutes (time excluding rest and warm up)
  Initial intensity = 3.2 km per hour and slope at 0% Walking until pain 3/5, then stop until pain completely subsides.Resume of walking as soon as possible.
  Increase :
  Week 1: if the walking is possible during 8 minutes, increase of the slope of 0.5% in each training until 10% Week 2 :if the walking is possible during 8 minutes, increase of the speed 0.2 mile per hour until 3 mph Week 3 :if the walking is possible during 8 minutes, increase of the slope 2% at each training until 15% Week 4 : if the walking is possible during 8 minutes, increase the speed 0.2mph at each training as long as it is possible.
  Arms: conventional rehabilitation program

SUMMARY:
Rehabilitation is the first intention treatment of peripheral arterial disease (PAD) with claudication. Initially proposed in the sixty's, rehabilitation programs dedicated to patients with PAD have recently been proved effective and defined in many guidelines. Supervised walking training on treadmill is recommended. Usually patients walk up to a mild or moderate pain (evaluated at 3 or 4 on the claudication pain scale; maximum pain =5), then stop until pain completely subsides and walk again .

The Artex study assesses the efficacy of a fractionated mode of training avoiding pain by alternating short sequences of intensive training and active recovery (without rest).

DETAILED DESCRIPTION:
Fractionated mode of training with active recovery has been proved effective in sport training as well as in Cardiac rehabilitation. We hypothesized it might be also interesting in the rehabilitation of patients with a peripheral arterial disease. The active recovery period might magnified the beneficial effect of a short intensive training.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male/female) between 18 and 80 years
* Patient with Fontaine stage II PAD confirmed by clinic, duplex ultrasound and ankle-to-brachial systolic blood pressure index
* Cardiac status compatible with an intensive gait rehabilitation (checked by a consultation with a cardiologist, including interview, clinical examination, electrocardiograph, and effort test on ergocycle).
* Volunteer to take part in the study, having sign the consent form after receiving sufficient information and the information leaflet
* Person affiliated to social security or the recipient of a similar scheme

Not Inclusion Criteria:

* Exercise tolerance limited by other factors than claudication (eg, coronary artery disease, dyspnea, poorly controlled blood pressure
* walking limited by other pathology
* osteoarticular lower limbs pathology
* abdominal aortic aneurysm > 4 cm
* pseudo-flu-like feverish syndromes in evolution (myocarditis or pericarditis)
* Person deprived of liberty by a legal or administrative decision, person under legal protection
* Person currently participating in a clinical trial or having taken part in a clinical trial in the month preceding inclusion
* Patient presenting with a history of mental or psychiatric illness or any other factor restricting his/her ability to participate in an informed manner and in compliance with the protocol

Exclusion Criteria:

Impossibility to perform protocol whatever reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intensive Rehabilitation in Peripheral Arterial Disease with Claudication: effects of a treadmill training with active recovery | Between day 0 and day 28
  Change in walking distance between day 0 and day 28, measured on a graded treadmill test

SECONDARY OUTCOMES:
Determine vascular and respiratory parameters which participate to improve the walking abilities after rehabilitation. | Between day 0 and day 28
  * Change in walking distance between day 0 and day 28, measured with the 6 MWT and the Strandness test.
  * Measure of ABI(Ankle-to- Brachial systolic blood pressure Index) and recovery time
  * Measure of the transcutaneous oxygen pression
  * Measure of the maximal cardiac frequency
  * Measure of peak oxygen consumption and lactatemy
Determine vascular and respiratory parameters which participate to improve the walking abilities after rehabilitation. | Between day 0 and day 28
  * Measure of ABI(Ankle-to- Brachial systolic blood pressure Index) and recovery time
  * Measure of the transcutaneous oxygen pression
  * Measure of the maximal cardiac frequency
  * Measure of peak oxygen consumption and lactatemy
One year follow-up | one year
  All patients included are invited to be assessed at a one year. Interview, Clinical Examination, and Assessemnts are performed in day hospital (half a day).
  Criteria are:
  Patients 'satisfaction about protocole using an ad hoc ordinal scale Medical and duplex scan examinations Vascular risk factors and comorbidities Occurence of any medical event during the year Changes in WIQ and HADS changes in walking distance at the Graduated Treadmill Test.
Reproducibility test of the walking graduated treadmill | Day 0 et day 1
  The fifteen last patients are invited to perform the consecutive graduated treadmill test on day 0 et day 1. Reproducibility of the walking distance assess by this novel test is quantified.

OTHER OUTCOMES:
Handicap and Depression measures | Between day 0 and day 28
  * Walking Impairment Questionary WIQ
  * Hospital Anxiety and Depression Scale HADS

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice VILLEMUR, MD, Principal Investigator — Unité de rééducation vasculaire - Clinique médecine physique de rééducation - CHU Grenoble - Hôpital Sud; Dominic Perennou, MD, PhD, Study Chair — Rehabilitation Department, Universitary Hospital Grenoble
Locations (1):
- CHU Grenoble - Hôpital Sud - Clinique médecine physique de rééducation, Échirolles, France

REFERENCES:
- [Background] Villemur B, Marquer A, Gailledrat E, Benetreau C, Bucci B, Evra V, Rabeau V, De Angelis MP, Bouchet JY, Carpentier P, Perennou D. New rehabilitation program for intermittent claudication: Interval training with active recovery: pilot study. Ann Phys Rehabil Med. 2011 Jul;54(5):275-81. doi: 10.1016/j.rehab.2011.05.003. Epub 2011 Jun 12. English, French. PMID 21704582
- [Background] Tisi PV, Hulse M, Chulakadabba A, Gosling P, Shearman CP. Exercise training for intermittent claudication: does it adversely affect biochemical markers of the exercise-induced inflammatory response? Eur J Vasc Endovasc Surg. 1997 Nov;14(5):344-50. doi: 10.1016/s1078-5884(97)80283-3. PMID 9413374
- [Background] Strandness DE Jr. Exercise testing in the evaluation of patients undergoint direct arterial surgery. J Cardiovasc Surg (Torino). 1970 May-Jun;11(3):192-200. No abstract available. PMID 5470199
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Nicolai SP, Viechtbauer W, Kruidenier LM, Candel MJ, Prins MH, Teijink JA. Reliability of treadmill testing in peripheral arterial disease: a meta-regression analysis. J Vasc Surg. 2009 Aug;50(2):322-9. doi: 10.1016/j.jvs.2009.01.042. PMID 19631868
- [Background] Meijer WT, Hoes AW, Rutgers D, Bots ML, Hofman A, Grobbee DE. Peripheral arterial disease in the elderly: The Rotterdam Study. Arterioscler Thromb Vasc Biol. 1998 Feb;18(2):185-92. doi: 10.1161/01.atv.18.2.185. PMID 9484982
- [Background] McDermott MM, Ades P, Guralnik JM, Dyer A, Ferrucci L, Liu K, Nelson M, Lloyd-Jones D, Van Horn L, Garside D, Kibbe M, Domanchuk K, Stein JH, Liao Y, Tao H, Green D, Pearce WH, Schneider JR, McPherson D, Laing ST, McCarthy WJ, Shroff A, Criqui MH. Treadmill exercise and resistance training in patients with peripheral arterial disease with and without intermittent claudication: a randomized controlled trial. JAMA. 2009 Jan 14;301(2):165-74. doi: 10.1001/jama.2008.962. PMID 19141764
- [Background] Le Faucheur A, Abraham P, Jaquinandi V, Bouye P, Saumet JL, Noury-Desvaux B. Measurement of walking distance and speed in patients with peripheral arterial disease: a novel method using a global positioning system. Circulation. 2008 Feb 19;117(7):897-904. doi: 10.1161/CIRCULATIONAHA.107.725994. Epub 2008 Feb 4. PMID 18250268
- [Background] Lechat P, Priollet P. [Prevention of major ischemic events in lower limb arterial disease: does aspirin play a role?]. J Mal Vasc. 2006 Jul;31(3):129-34. doi: 10.1016/s0398-0499(06)76531-3. French. PMID 16840949
- [Background] Kruidenier LM, Nicolai SP, Hendriks EJ, Bollen EC, Prins MH, Teijink JA. Supervised exercise therapy for intermittent claudication in daily practice. J Vasc Surg. 2009 Feb;49(2):363-70. doi: 10.1016/j.jvs.2008.09.042. Epub 2008 Nov 22. PMID 19028059
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Harvey SB, Hotopf M, Overland S, Mykletun A. Physical activity and common mental disorders. Br J Psychiatry. 2010 Nov;197(5):357-64. doi: 10.1192/bjp.bp.109.075176. PMID 21037212
- [Background] Montgomery PS, Gardner AW. The clinical utility of a six-minute walk test in peripheral arterial occlusive disease patients. J Am Geriatr Soc. 1998 Jun;46(6):706-11. doi: 10.1111/j.1532-5415.1998.tb03804.x. PMID 9625185
- [Background] Gardner AW, Skinner JS, Smith LK. Effects of handrail support on claudication and hemodynamic responses to single-stage and progressive treadmill protocols in peripheral vascular occlusive disease. Am J Cardiol. 1991 Jul 1;68(1):99-105. doi: 10.1016/0002-9149(91)90719-2. PMID 2058566
- [Background] Gardner AW, Katzel LI, Sorkin JD, Goldberg AP. Effects of long-term exercise rehabilitation on claudication distances in patients with peripheral arterial disease: a randomized controlled trial. J Cardiopulm Rehabil. 2002 May-Jun;22(3):192-8. doi: 10.1097/00008483-200205000-00011. PMID 12042688
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Gardner AW, Skinner JS, Cantwell BW, Smith LK. Progressive vs single-stage treadmill tests for evaluation of claudication. Med Sci Sports Exerc. 1991 Apr;23(4):402-8. PMID 2056896
- [Background] Gardner AW, Poehlman ET. Assessment of free-living daily physical activity in older claudicants: validation against the doubly labeled water technique. J Gerontol A Biol Sci Med Sci. 1998 Jul;53(4):M275-80. doi: 10.1093/gerona/53a.4.m275. PMID 18314566
- [Background] Fife CE, Smart DR, Sheffield PJ, Hopf HW, Hawkins G, Clarke D. Transcutaneous oximetry in clinical practice: consensus statements from an expert panel based on evidence. Undersea Hyperb Med. 2009 Jan-Feb;36(1):43-53. PMID 19341127
- [Background] Crowther RG, Spinks WL, Leicht AS, Quigley F, Golledge J. Relationship between temporal-spatial gait parameters, gait kinematics, walking performance, exercise capacity, and physical activity level in peripheral arterial disease. J Vasc Surg. 2007 Jun;45(6):1172-8. doi: 10.1016/j.jvs.2007.01.060. PMID 17543681
- [Background] Bruce RA, Kusumi F, Hosmer D. Maximal oxygen intake and nomographic assessment of functional aerobic impairment in cardiovascular disease. Am Heart J. 1973 Apr;85(4):546-62. doi: 10.1016/0002-8703(73)90502-4. No abstract available. PMID 4632004
- [Background] Bronas UG, Hirsch AT, Murphy T, Badenhop D, Collins TC, Ehrman JK, Ershow AG, Lewis B, Treat-Jacobson DJ, Walsh ME, Oldenburg N, Regensteiner JG; CLEVER Research Group. Design of the multicenter standardized supervised exercise training intervention for the claudication: exercise vs endoluminal revascularization (CLEVER) study. Vasc Med. 2009 Nov;14(4):313-21. doi: 10.1177/1358863X09102295. PMID 19808716
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Baker JD, Dix DE. Variability of Doppler ankle pressures with arterial occlusive disease: an evaluation of ankle index and brachial-ankle pressure gradient. Surgery. 1981 Jan;89(1):134-7. PMID 7466604
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Derived] Villemur B, Thoreau V, Guinot M, Gailledrat E, Evra V, Vermorel C, Foote A, Carpentier P, Bosson JL, Perennou D. Short interval or continuous training programs to improve walking distance for intermittent claudication: Pilot study. Ann Phys Rehabil Med. 2020 Nov;63(6):466-473. doi: 10.1016/j.rehab.2020.03.004. Epub 2020 Apr 6. PMID 32272287